CLINICAL TRIAL: NCT00273143
Title: Kinetics of Cytomegalovirus (CMV) Replication and CMV-specific Immune Reconstitution After Hematopoietic Stem Cell Transplantation.
Brief Title: A Trial to Study How the Body Fights Off Cytomegalovirus (CMV) in Hematopoietic Transplant Recipients.
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Other Study IDs: 1052-05
Record Dates: First submitted 2006-01-06; First posted 2006-01-09 (Estimated); Last update posted 2011-05-24 (Estimated); Status verified 2011-05

CONDITIONS: Cytomegalovirus Infection
MeSH Terms: conditions — Cytomegalovirus Infections

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This study is being done to determine how the body fights off a common virus known as Cytomegalovirus (CMV). CMV is a virus that commonly infects humans and causes disease in patients with compromised immune function such as those who receive organ and tissue transplant. By knowing how the human body responds to the infection, researchers will be able to develop better methods on how to prevent this infection.

DETAILED DESCRIPTION:
This study is looking at the CMV virus in Hematopoietic stem cell donors and recipients. In the donor population, the study is looking at the participants blood to see if they contain cells that are active against the virus. Information about the donor will be obtained through an interview and through review of medical records. A blood sample will be drawn at the time of the donor's evaluation, which will take place in conjunction with the regular blood tests that are ordered. Participants of the study who are donors will only be involved in the study at the time of blood collection.

Participants who will be receiving hematopoietic stem cell transplantation will have data collected through an interview and review of medical records. Participants will have blood drawn prior to transplant, weekly for 12 weeks and then monthly for three months following transplant. In addition, if CMV disease develops during this period of time, blood will be drawn till the participant is cured for the disease. All blood draws for thes study will take place in conjunction with the regular routine blood work. Participants will be in the study for one year after transplant.

ELIGIBILITY:
Participants who will be undergoing blood marrow or stem cell transplant and donors that are 18 years of age or older, may be eligible to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: rticipants who will be undergoing blood marrow or stem cell transplant and donors that are 18 years of age or older, may be eligible to participate in this study.
Sampling Method: Probability Sample
Enrollment: 50
Dates: Start 2005-05; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
To characterize the kinetics of CMV-specific immunity after HSCT.
To characterize the kinetics of CMV replication after HSCT.
To assess the degree of Epstein-Barr virus (EBV), human herpesvirus (HHV)-6 and HHV-7 replication after HSCT.

CONTACTS AND LOCATIONS:
Overall Officials: Raymund R. Razonable, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States